CLINICAL TRIAL: NCT06906185
Title: Adaptation and Examination of a Trauma-informed Intervention for Pregnant Veterans (CDA 22-135)
Brief Title: Adaptation and Examination of a Trauma-informed Intervention for Pregnant Veterans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CDX 25-002; IK2HX003681-01A2 (NIH)
Record Dates: First submitted 2025-03-18; First posted 2025-04-02 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Trauma-related Mental Health Symptoms
Keywords: Anxiety; Depression; PTSD; Pregnant Veteran; Reproductive Mental Health
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: During Aim 2, Veterans are randomly assigned (1:1 using a random number generated table) to the active (Calm Moms-V) or control (care as usual in VHA) condition.
  Aim 1 and Aim 3 do not involve a clinical trial or randomization.
Masking Description: N/A - masking not used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): The active condition will be the Calm Moms-V treatment.
  Interventions: Behavioral: Calm Moms-V
- Control (Active Comparator): The control condition will be care as usual in VHA.
  Interventions: Behavioral: Care As Usual

INTERVENTIONS:
Behavioral: Calm Moms-V — Calm Moms-V is the trauma-informed treatment developed and refined by the PI and being tested in the current study. Calm Moms-V is an online treatment program for trauma-exposed pregnant Veterans designed to target anxiety, stress, low mood, and trauma-related symptoms using empirically supported CBT techniques. Calm Moms-V includes four sessions and a booster session closer to delivery/postpartum. Sessions 1-4 are designed to be completed across four weeks (one session delivered each week). Each session is self-paced and designed to take approximately 45 minutes to complete.
  Arms: Active
Behavioral: Care As Usual — The control condition will be Care As Usual (CAU). CAU at SLVHCS involves participation in available services chosen by the patient with input from their providers. Further, for all pregnant Veterans that use VHA maternity benefits, CAU includes routine phone calls (throughout pregnancy and up to one-year postpartum) conducted by the site MCC to coordinate maternity benefits, facilitate additional services, and arrange for specific supplies (e.g., breast pump). Further, the SLVHCS MCC mails each pregnant Veteran enrolled in VHA a "welcome packet" that includes national, local, and VHA MH and physical health resources that may be useful to them during the perinatal period. Veterans in the CAU condition will be assessed at the same intervals as those in the active condition.
  Arms: Control

SUMMARY:
The current proposal aims to refine and examine an intervention called Calm Moms. Calm Moms is a web-based treatment program designed to reduce anxiety, stress, and low mood symptoms among pregnant Veterans with a history of trauma exposure. Its contents are based on empirically supported cognitive behavioral therapy (CBT) techniques shown to be effective in reducing these symptoms. Further, the Calm Moms program is tailored towards the unique concerns of pregnant women and incorporates information on how to cope with and reduce the impact of trauma. Calm Moms may benefit pregnant Veterans by reducing their anxiety, stress, and low mood symptoms. Additionally, pregnant Veterans who engage in Calm Moms may have improved functioning, reduced impairment during pregnancy, and show increased interest and engagement with additional mental health care. The current proposal also aims to collect information regarding implementation of Calm Moms at additional sites, which will allow Calm Moms to impact a larger group of pregnant Veterans.

DETAILED DESCRIPTION:
Background: Trauma exposure and subsequent mental health symptoms are exceptionally common among pregnant Veterans and associated with a variety of negative perinatal outcomes (e.g., postpartum depression, gestational diabetes, low birth weight). The mechanism linking trauma exposure and poor perinatal outcomes is elevated anxiety, stress, and low mood during pregnancy. Thus, treatments designed to target these symptoms among trauma-exposed pregnant Veterans are critical. The Veterans Health Administration (VHA) has started to address this need, but the available treatments are not sufficient because they do not address two common symptoms of trauma exposure (i.e., anxiety and stress) or mental health symptoms during pregnancy. Further, pregnant Veterans with a trauma history report myriad barriers to engaging in mental health treatment (e.g., stigma, accessibility, and availability). Calm Moms-V is a treatment program that directly addresses the gaps in care and barriers to treatment for this vulnerable population. Calm Moms-V is an online treatment program rooted in empirically supported cognitive behavioral therapy (CBT) techniques shown to be effective in reducing anxiety and stress and improving mood. Calm Moms-V was adapted from the original Calm Moms program (based on Veteran stakeholder feedback) and now includes four weekly sessions and a booster session close to delivery/postpartum. The current study will build on this work by examining the resulting Calm Moms-V among pregnant Veterans.

Significance: Although a small proportion of the Veteran population, pregnant Veterans are especially vulnerable because they (1) have often recently transitioned from Active Duty, (2) carry a heavy burden of trauma and mental health symptoms, (3) often have partners still on Active Duty, and (4) face fragmented care because obstetrics services must be provided by community providers. Calm Moms-V is an accessible, low-cost, and evidence-based treatment program. Pregnant Veterans who engage in Calm Moms-V may (1) experience a reduction in anxiety, stress, and low mood during pregnancy, (2) have improved functioning and reduced impairment during pregnancy, and (3) show interest and engagement with VHA mental health care.

Innovation/Impact: Trauma-exposed pregnant Veterans have low mental health engagement and report a disinterest in traditional trauma-focused treatment; however, they have among the worst perinatal outcomes, in part due to elevated mental health symptoms. Calm Moms-V will directly address these gaps by providing a program that may reduce anxiety, stress, and low mood symptoms and enhance engagement in mental health treatment.

Specific Aims: The current study aims to: (1) Collect feedback on Veteran experience with Calm Moms-V and make final refinements, (2) Conduct a pilot acceptability and feasibility trial of Calm Moms-V at SLVHCS, and (3) Examine barriers and facilitators to implementation of Calm Moms-V at additional sites.

Methodology: The current study will utilize a mixed-methods approach targeting pregnant Veterans and key VHA stakeholders.

Next Steps/Implementation: This research has the long-term potential to make trauma-informed mental health care readily available for all pregnant Veterans. Although the implementation and dissemination implications of Calm Moms-V are nascent, Calm Moms-V may be useful in a stepped-care framework or as a way to connect pregnant Veterans with additional mental health care. Data from this study will be used to inform additional research aimed at examining the broad implementation of Calm Moms-V in VHA. Further, in collaboration with the study partners, the investigators will work to disseminate results from this study and treatment materials through various local and national outlets.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant (any trimester)
* Endorse a DSM-5-TR Criterion A traumatic event as indexed by the trauma exposure portion of the PTSD screen for primary care (PC-PTSD-5)
* Endorse clinically elevated anxiety (as indexed by a total score of > 3 on the GAD-2) or depression symptoms (as indexed by a total score of > 3 on the PHQ-2)
* Able to participate in an online intervention (i.e., have internet and smartphone, tablet, or computer access)

Of note, pregnant Veterans will still be eligible if they are in concurrent psychotherapy and/or using psychotropic medications.

Exclusion Criteria:

* Evidence of a significant mental illness that would impede completion of the intervention

  * (i.e., active psychosis, uncontrolled bipolar disorder, a severe alcohol/substance use disorder, or suicidal ideation or behavior that requires immediate hospitalization or treatment)

Evidence of a significant mental illness will be determined via pre-enrollment chart review.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2028-09-29 (Estimated); Study Completion 2030-03-29 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM) | Aim 2 at one-month follow-up and at three-month follow-up.
  The Acceptability of Intervention Measure (AIM) is a brief self-report measures designed to assess the extent to which an intervention is acceptable. Scores range from 8 to 40 with higher scores indicating greater acceptability (better outcome = high acceptability). The AIM is psychometrically sound and have been validated in previous research. The AIM will be administered to Veterans randomized to Calm Moms-V during the one-month and three-month follow-up assessments.
Feasibility of Intervention Measure (FIM) | Aim 2 at one-month follow-up and at three-month follow-up.
  The Feasibility of Intervention Measure (FIM) is a brief self-report measures designed to assess the extent to which an intervention is feasible. Scores range from 8 to 40 with higher scores indicating greater feasibility (better outcome = high feasibility). The FIM is psychometrically sound and has been validated in previous research. The FIM will be administered to Veterans randomized to Calm Moms-V during the one-month and three-month follow-up assessments.

SECONDARY OUTCOMES:
Work and Social Adjustment Scale (WSAS) | Aim 2 at all assessment timepoints (baseline, one-month follow-up, two-month follow-up, and three-month follow-up).
  The Work and Social Adjustment Scale (WSAS) will be used to assess functional impairment due to mental health difficulties over time. Scores range from 0 to 40 with higher scores indicating greater functional impairment (worse outcome = high scores or increased functional impairment). The WSAS is psychometrically sound and has been validated in previous research. The WSAS will be administered at all assessment timepoints (baseline, one-month follow-up, two-month follow-up, and three-month follow-up) to examine changes in functioning and impairment over time.

OTHER OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | Aim 2 at all assessment timepoints (baseline, one-month follow-up, two-month follow-up, and three-month follow-up).
  The Generalized Anxiety Disorder-7 (GAD-7) will be used to assess anxiety symptoms over time. Scores range from 0 to 21 with higher scores indicating greater anxiety symptoms (worse outcome = high score or higher anxiety symptoms). The GAD-7 is psychometrically sound and has been validated in previous research. The GAD-7 will be administered at all assessment timepoints (baseline, one-month follow-up, two-month follow-up, and three-month follow-up) to examine changes in anxiety over time.
Patient Health Questionnaire-9 (PHQ-9) | Aim 2 at all assessment timepoints (baseline, one-month follow-up, two-month follow-up, and three-month follow-up).
  The Patient Health Questionnaire-9 (PHQ-9) will be used to assess depression symptoms over time. Scores range from 0 to 27 with higher scores indicating greater depression symptoms (worse outcome = high score or higher depression symptoms). The PHQ-9 is psychometrically sound and has been validated in previous research. The PHQ-9 will be administered at all assessment timepoints (baseline, one-month follow-up, two-month follow-up, and three-month follow-up) to examine changes in depression over time.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Shapiro, PhD MS, Principal Investigator — Southeast Louisiana Veterans Health Care System, New Orleans, LA
Locations (1):
- Southeast Louisiana Veterans Health Care System, New Orleans, LA, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No